CLINICAL TRIAL: NCT07317557
Title: Mechanisms of Remote Ischemic Conditioning in Preventing and Treating Cognitive Impairment in Cerebral Small Vessel Disease
Brief Title: Remote Ischemic Conditioning for Cognitive Impairment in Cerebral Small Vessel Disease
Acronym: RIC-CSVD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-KY142-01; 82402970 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-12-08; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Small Vessel Disease; Cognitive Impairment
Keywords: cerebral small vessel disease; cognitive impairment; remote ischemic conditioning; white matter hyperintensities; EEG functional connectivity
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental): Remote ischemic conditioning plus standard medical therapy.
  Interventions: Device: Remote ischemic conditioning using IPC-906 device
- Sham remote ischemic conditioning (Sham Comparator): Sham remote ischemic conditioning plus standard medical therapy
  Interventions: Device: Sham remote ischemic conditioning using IPC-906 device

INTERVENTIONS:
Device: Remote ischemic conditioning using IPC-906 device — A pneumatic cuff is placed on one upper limb and inflated to 200 mmHg for 5 minutes followed by 5 minutes of reperfusion, repeated for 5 cycles (total 45 minutes) per session, twice daily for 90 days, in addition to standard medical therapy.
  Arms: Remote ischemic conditioning
Device: Sham remote ischemic conditioning using IPC-906 device — The same cuff procedure is applied, but cuff pressure is set at 60 mmHg, which does not induce ischemia. The schedule is identical: 5 minutes inflation and 5 minutes reperfusion, 5 cycles (45 minutes) per session, twice daily for 90 days, in addition to standard medical therapy.
  Arms: Sham remote ischemic conditioning

SUMMARY:
This randomized, double-blind, sham-controlled trial aims to evaluate the effect of remote ischemic conditioning (RIC) on cognitive function in patients with cerebral small vessel disease-related mild cognitive impairment. Forty eligible participants will be randomized 1:1 to receive either RIC or sham RIC twice daily for 90 days in addition to standard medical therapy. The primary outcome is the change in Montreal Cognitive Assessment (MoCA) score from baseline to 90 days. Secondary outcomes include changes in white matter hyperintensity burden and diffusion tensor imaging metrics on MRI, EEG functional connectivity, and activities of daily living.

DETAILED DESCRIPTION:
Cerebral small vessel disease (CSVD) is a leading cause of vascular cognitive impairment, characterized by white matter hyperintensities, lacunes, and microbleeds on MRI. Current treatment options for CSVD-related cognitive impairment are limited, and there is a critical need for safe, noninvasive interventions that can improve cognitive function and delay disease progression.

Remote ischemic conditioning (RIC) is a noninvasive, low-cost procedure induced by intermittent cuff inflation on a limb to produce brief episodes of ischemia and reperfusion. Experimental and clinical studies suggest that RIC can improve cerebral perfusion, protect the neurovascular unit, and modulate inflammatory and endothelial pathways, making it a promising strategy for CSVD.

In this single-center, randomized, double-blind, sham-controlled trial, we will enroll 40 patients with CSVD-related mild cognitive impairment. Participants will be randomized to receive either RIC (cuff inflation to 200 mmHg for 5 minutes followed by 5 minutes of reperfusion, 5 cycles per session) or sham RIC (cuff inflation to 60 mmHg, 5 cycles per session). The intervention will be administered twice daily for 90 days, in addition to standard medical therapy.

Cognitive function will be assessed by the Montreal Cognitive Assessment (MoCA). MRI will be used to quantify white matter hyperintensities and diffusion tensor imaging parameters, and EEG will be used to evaluate functional connectivity. Activities of daily living and safety outcomes will also be recorded. This study will provide clinical and mechanistic evidence on whether RIC can prevent or ameliorate cognitive impairment in patients with CSVD.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years.
* Diagnosis of cerebral small vessel disease according to the Chinese Guidelines for the Diagnosis and Treatment of Cerebral Small Vessel Disease (2020).
* Mild cognitive impairment with a Montreal Cognitive Assessment (MoCA) score of 18-25.
* The patient or a legally authorized representative is able and willing to sign written informed consent.

Exclusion Criteria:

* Any condition that is unsuitable for remote ischemic conditioning, including soft tissue injury, limb deformity or vascular injury in the upper limb, bleeding disorders, or systolic blood pressure > 200 mmHg.
* History or presence of neurological or psychiatric disorders that may interfere with participation or outcome assessment, such as other cerebrovascular diseases, Parkinson's disease, or major depressive disorder.
* Current or past severe systemic diseases deemed inappropriate for the study by the investigator, including but not limited to severe cardiovascular diseases (e.g., congestive heart failure, severe arrhythmia, myocardial infarction), severe hepatic diseases (e.g., cirrhosis), severe renal diseases (e.g., requiring hemodialysis or peritoneal dialysis), hematologic diseases with bleeding tendency (e.g., hemophilia), poorly controlled diabetes (blood glucose > 16.8 mmol/L or < 2.8 mmol/L) or with severe complications, active or uncontrolled systemic autoimmune diseases or primary/secondary immunodeficiency, or malignancy.
* Laboratory abnormalities, including absolute neutrophil count < 1.5 × 10⁹/L, platelet count < 100 × 10⁹/L, hemoglobin < 90 g/L, AST or ALT > 2.5 × upper limit of normal (ULN), total bilirubin > 1.5 × ULN, or serum creatinine > 1.5 × ULN.
* Coagulation abnormalities, including for patients not on anticoagulant/antithrombotic therapy: INR > 1.7 or APTT > 1.25 × ULN; and for patients on anticoagulant/antithrombotic therapy: INR > 3.0 or APTT > 1.5 × ULN.
* Positive tests for hepatitis B with detectable HBV-DNA, or positive serology for hepatitis C, syphilis (TPAb/RPR), or HIV.
* Pregnant or breastfeeding women.
* Contraindications to MRI (e.g., pacemaker or other metallic implants, severe claustrophobia).
* Participation in another clinical trial within 3 months prior to enrollment.
* Severe trauma or major surgery within 3 months before remote ischemic conditioning, or planned surgery during the study period (except minor procedures and laparoscopic procedures performed within 4 weeks before baseline).
* History of substance abuse or alcoholism within 1 year prior to enrollment.
* Any other condition that may increase risk or interfere with the interpretation of study results, as judged by the investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) score from baseline to 90 days. | Baseline and 90 days after randomization.
  The primary endpoint is the difference in mean MoCA score change from baseline to 90 days between the remote ischemic conditioning group and the sham group.

SECONDARY OUTCOMES:
Change in total white matter hyperintensity (WMH) volume on brain MRI (milliliters). | Baseline and 90 days.
  Total WMH volume (mL) will be quantified on 3D T2-FLAIR brain MRI using semi-automated volumetric segmentation and normalized to intracranial volume. The outcome is the change in total WMH volume from baseline to 90 days between the two groups.
Change in mean diffusivity (MD) of cerebral white matter on diffusion tensor MRI (×10-³ mm²/s). | Baseline and 90 days.
  Mean diffusivity (×10-³ mm²/s) will be calculated from diffusion tensor imaging in predefined cerebral white matter regions of interest. The outcome is the change in MD from baseline to 90 days between the two groups.
Change in fractional anisotropy (FA) of cerebral white matter on diffusion tensor MRI. | Baseline and 90 days.
  Fractional anisotropy values in predefined cerebral white matter regions will be derived from diffusion tensor imaging. The outcome is the change in FA from baseline to 90 days between the two groups.
Change in axial diffusivity (AD) of cerebral white matter on diffusion tensor MRI (×10-³ mm²/s). | Baseline and 90 days.
  Axial diffusivity (×10-³ mm²/s) in predefined cerebral white matter regions will be obtained from diffusion tensor imaging. The outcome is the change in AD from baseline to 90 days between the two groups.
Change in radial diffusivity (RD) of cerebral white matter on diffusion tensor MRI (×10-³ mm²/s). | Baseline and 90 days.
  Radial diffusivity (×10-³ mm²/s) in predefined cerebral white matter regions will be obtained from diffusion tensor imaging. The outcome is the change in RD from baseline to 90 days between the two groups.
Change in EEG global functional connectivity (graph-theoretical global efficiency index). | Baseline and 90 days.
  Weighted functional connectivity matrices will be constructed from resting-state EEG signals, and graph-theoretical global efficiency (dimensionless) will be calculated as a summary index of whole-brain functional connectivity. The outcome is the change in global efficiency from baseline to 90 days between the two groups.
Change in Activities of Daily Living (ADL) scale score. | Baseline and 90 days.
  The Activities of Daily Living Scale (ADL) is a [[X-item]] questionnaire assessing basic daily self-care abilities. Each item is scored from [[A]] to [[B]] points, yielding a total score ranging from [[0]] to [[100]] points. Higher scores indicate worse activities of daily living (greater functional impairment). The outcome is the change in ADL total score from baseline to 90 days between the two groups.
Incidence of adverse events related to remote ischemic conditioning. | Baseline to 90 days.
  Including skin petechiae, bruising, limb discomfort or numbness, and any serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyin Wang, MD, Principal Investigator — Department of Neurology, Nanjing Brain Hospital
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data (IPD) from this trial with external researchers. De-identified, aggregate study results will be reported in publications and presentations in accordance with institutional and national regulations.